CLINICAL TRIAL: NCT01191463
Title: The Efficacy of a Local Vitamin-C Rich Fruit (Guava) in Improving Iron Absorption From Mungbean Based Meals in Indian Children (6-10 Years)
Brief Title: The Efficacy of a Local Vitamin-C Rich Fruit (Guava) in Improving Iron Absorption From Mungbean Based Meals and Its Effect on Iron Status of Rural Indian Children (6-10 Years)
Acronym: MUGUST_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: CCS Haryana Agricultural University Hisar, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MUGUST_2
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Iron Deficiency; Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mung Bean Meals and Guava fruit (Experimental): Subject in this group will receive, a lunch meal based on 50g of Mung beans together with a local, Vitamin C rich fruit (Guava)
  Interventions: Other: Mung Bean Meal; Other: Guava
- Mung Bean (Active Comparator): Subjects in this group will receive a lunch meal based on 50g mung beans but without any vitamin C source.
  Interventions: Other: Mung Bean Meal
- School feeding program (No Intervention): Subjects in this arm, will receive the regular school feeding program as provided by the school authorities

INTERVENTIONS:
Other: Mung Bean Meal — 50g mung beans will be cooked to a curry with oil, spices and small amounts of vegetables.
  Arms: Mung Bean; Mung Bean Meals and Guava fruit
Other: Guava — A fresh Guava fruit will be provided raw (approx 100g fresh weight)
  Arms: Mung Bean Meals and Guava fruit

SUMMARY:
Iron deficiency is estimated to affect about one fifth of the world's population, and women and children are among the most severely affected. Evidence is mounting that iron deficiency anemia adversely affects brain development with measurable effects on children's behavior, motor development and cognition. In Hisar district of Haryana state, north- India, 58% of school age children (6-10 years) are anemic, 49 % are iron deficient whereas 40 % have been found to be anemic due to iron deficiency. Iron bioavailability calculated using algorithms in regional diets ranged from 3.2 to 4.6 percent. Mungbean (Vigna radiata L.) is the third most important legume crop of India. It is a high potential legume crop with 4-8 mg of iron and known as a nutritious and healthy legume. Ascorbic acid is a potent enhancer of iron absorption in humans which can counteract the inhibitory effect of phytic acid and polyphenols. Guava is a popular and easily available fruit for this community having 200- 300 mg/100g of ascorbic acid. We will conduct a randomised controlled trial in school age children (6-10 years) in Haryana state of India, to determine the efficacy of local vitamin-C rich fruit guava with mungbean based meal on iron status of rural Indian children.

Objective: To assess the effect of mungbean based test meal on iron status (as body iron stores, defined and calculated by the ratio of serum ferritin and serum transferrin receptor) of school age children (6-10 years) with and without the consumption of guava, a vitamin C rich fruit, in a school feeding program for seven months.

Study population: Three hundred school children aged between 6-10 years will be recruited from two government school of Mangali village situated in Hisar district of Haryana state.

Study design: This intervention study will be carried out in a randomized controlled design. Main study parameters/endpoints: Primary outcome will be the measurement of body iron stores (mg/kg of body weight) based on the ratio of serum transferrin receptor to serum ferritin.

DETAILED DESCRIPTION:
Primary Objective To measure the effect of mungbean based test meal on iron status (defined by body iron stores, calculated as the ratio of ferritin and serum transferrin receptor) of school age children (6-10 years) with and without the consumption of guava, a vitamin C rich fruit, distributing in school feeding program for seven months.

Three weeks before the trial available children (6-10 years) in selected schools will be screened for eligibility of the study on the basis of medical health questionnaire. Deworming will be done at least 20 days before the start the feeding trial with a single dose of Albendazole (400 mg), that will be given again after three months. These 300 children will be assigned to three groups (100 children each group). Group-1 will be served with the normal school feeding program (SFP) meal (see annexure-1) and this group will also serve as control group for the study. Group-2 will be served with mungbean test meal (see annexure-2) and group-3 will be served with guava fruit in addition of mungbean test meal. Meals to all children will be provided for six days in a week up to seven months. All meals will be served at mid morning (11.00 am to 11.30 am). Effect of intervention will be assessed in terms of iron status of children.

This study will be carried out in two government schools of Mangali village belong to Hisar-1 block of Hisar district Haryana state with the close supervision of Chaudhary Charan Singh Haryana Agriculture University, Hisar.

Children having severe anemia (Hb <7.0 g/dl) will be excluded from the trial and referred for medical treatment.

Subjects will be recruited that comply with the following criteria:

* School children (6-10) years of age,
* enrolled in selected primary schools,
* Informed consent obtained from at least one parent or guardian,
* Children should be apparently healthy; i.e. have no pre-existing medical conditions or be receiving chronic medication,
* Should not be allergic / hypersensitive to any of the ingredients of the test meal, Should not consume mineral/vitamin supplements.
* If the child consume supplements he/she will be asked to stop taking the supplements two weeks before the study and during the study.

A total of two blood samples will be taken from the participants, one at the start of the study, and second at the end of the study. With each sampling 7ml blood will be taken by an experienced technician. Blood will always be drawn in the morning between 7.30 and 9.00am at particular school by the well trained technician. Hemoglobin in whole blood, serum ferritin (Sf), serum transferrin receptor (sTfR), serum CRP and AGP will be analysed to compare the iron status. Body iron stores will be calculated with the formula by Cook et. al. All analysis will be carried out at the same time for both samples of baseline and after intervention at St. John hospital, Bangalore. Therefore serum samples of baseline will be stored for seven months at - 800c temperature. The CV of intra-assays and inter-assays will be, monitored. Blood samples will not be destroyed after completion the study they will be kept for up to 5 years.

Iron status will be compared in children belonging to three different groups in pre and post conditions, using above mentioned iron status indicators. Height and weight of the children will also be measured at pre and post of the intervention study. The primary outcome of this study will be body iron stores calculated with the cook formula.

Secondary outcomes will be prevalence of iron deficiency, anaemia, and difference in haemoglobin concentration and plasma concentrations of ferritin, and soluble transferring receptor in the two treatment groups. Anemia will be defined as a hemoglobin concentration <11.5g/L and iron deficiency will be defined as an SF concentration <12µg/l. The cut-off for normal CRP and AGP are defined at <5mg/L and <1g/L(12), respectively. Anthropometric indices will be calculated using WHO (2006) (10) Child growth standards. Being stunted, underweight or wasted will be defined by Z score <-2SD for height-for-age, weight-for-age and weight-for-height respectively.

ELIGIBILITY:
Inclusion Criteria:

* School children (6-10) years of age
* Enrolled in selected primary schools
* Informed consent obtained from at least one parent or guardian
* Children should be apparently healthy; i.e. have no pre-existing medical conditions or be receiving chronic medication.
* Should not be allergic / hypersensitive to any of the ingredients of the test meal
* Should not consume mineral/vitamin supplements. If the child consume supplements he/she will be asked to stop taking the supplements two weeks before the study and during the study

Exclusion Criteria:

* Subjects with severe anemia (Hb=70 g/L)will be referred for treatement at the local health facility.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Body Iron Stores | Baseline (Start month=0), End of study (Month=7)
  Defined as the ration between serum ferritin and soluble serum transferrin recpetor Body iron stores are a sensitive measure of body iron balance and indicative of body iron changes.

SECONDARY OUTCOMES:
Prevalence of iron deficiency, Prevalence of Iron deficiency anemia | Begin (Month=0), End (Month=7)
  Anemia will be defined as a hemoglobin concentration <11.5g/L and iron deficiency will be defined as an SF concentration <12µg/l.

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Rani, PhD, Principal Investigator — Wageningen University, Haryana University
Locations (1):
- CCS Haryana Agricultural University, Hisar, Haryana State, India

REFERENCES:
- [Background] Rani, V., Brouwer, Inge., Khetarpaul, N., Zimmerman, M.B. (2009) Iron status and associated factors in rural school going children (5-8 years) of Haryana state, India., Abstract Book Wageningen Nutritional Sciences Forum March 4-6, 2009 European Journal of Clinical Nutrition, 63 (3S) Pp:20
- [Derived] Rani V, Moretti D, Khetarpaul N, Thankachan P, Zimmermann MB, Melse-Boonstra A, Brouwer ID. Vitamin C-Rich Guava Consumed with Mungbean Dal Reduces Anemia and Increases Hemoglobin but not Iron Stores: A Randomized Controlled Trial of Food-to-Food Fortification in Indian Children. J Nutr. 2024 Dec;154(12):3740-3748. doi: 10.1016/j.tjnut.2024.10.042. Epub 2024 Oct 30. PMID 39481541